CLINICAL TRIAL: NCT07031648
Title: The Effect Of Laughter Yoga And Pilates On Pregnancy Compliance, Anxiety And Prenatal Attachment In Pregnant Women Receiving Childbirth Preparation Training
Brief Title: The Effect of Laughter Yoga and Pilates on Pregnancy in Pregnant Women Receiving Childbirth Preparation Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Demet Guney, MSc., Research Assist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: Kastamonu
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prenatal Care
Keywords: pilates; Laughter Yoga; Anxiety; Prenatal Attachment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Type of Study: It is a randomized controlled experimental study and is planned based on the pre-test-post-test model
  Pregnant women randomly assigned to the Laughter Yoga and Pilates Group constitute the experimental group of the study.
  Only those who received planned training for pregnancy and postpartum constituted the control group of the study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laughter Yoga Group (Experimental): Giving information about the yoga of meeting and laughter, Obtaining written consent through the informed consent form, Pre-test will be applied in the first week Providing routine pregnancy school trainings by midwife trainers in the pregnancy school, Practicing laughter yoga 2 times a week for 4 weeks for a total of 8 sessions, Sessions should consist of a maximum of 15 people, A total of 45 minutes of laughter sessions for pregnant women, At the end of the fourth week, the final test will be administered
  Interventions: Other: Laughter Yoga Group
- Pilates Group (Experimental): Providing information about meeting and Pilates, Obtaining written consent through the informed consent form, Pre-test will be applied in the first week Providing routine pregnancy school trainings by midwife trainers in the pregnancy school, Performing a total of 8 sessions of pregnant pilates exercises for 4 weeks, 2 times a week, Sessions should consist of a maximum of 10 people, A total of 45 minutes of pilates exercise for pregnant women, At the end of the fourth week, the final test will be administered
  Interventions: Other: Pilates Group
- Education Group (Other): Providing information about the research, Obtaining written consent through the informed consent form, Pre-test will be applied in the first week Providing routine pregnancy school trainings by midwife trainers in the pregnancy school (pregnancy, postpartum care, baby care, breastfeeding, etc.) At the end of the fourth week, the final test will be administered
  Interventions: Other: Education Group

INTERVENTIONS:
Other: Laughter Yoga Group — iving information about the yoga of meeting and laughter, Obtaining written consent through the informed consent form, Pre-test will be applied in the first week Providing routine pregnancy school trainings by midwife trainers in the pregnancy school, P
  Arms: Laughter Yoga Group
Other: Pilates Group — Providing information about meetings and Pilates, Obtaining written consent through an informed consent form, Pre-test will be applied in the first week Providing routine pregnancy school trainings by midwife trainers in the pregnancy school, Doing a total of 8 sessions of pregnant pilates exercises for 4 weeks, 2 times a week, Sessions should consist of a maximum of 10 people, A total of 45 minutes of pilates exercise for pregnant women, At the end of the fourth week, the final test will be administered
  Arms: Pilates Group
Other: Education Group — Providing information about the research, Obtaining written consent through the informed consent form, Pre-test will be applied in the first week Providing routine pregnancy school trainings by midwife trainers in the pregnancy school (pregnancy, postpartum care, baby care, breastfeeding, etc.) At the end of the fourth week, the final test will be administered
  Arms: Education Group

SUMMARY:
The aim of the study was to determine the effect of laughter yoga and pilates on pregnancy adjustment, anxiety and prenatal attachment in pregnant women who received childbirth preparation training.

DETAILED DESCRIPTION:
Pregnancy, childbirth and the process of becoming a parent are important life events in women's lives. Since birth is an unpredictable and uncontrollable process, this process may be accompanied by stress, fear and anxiety from time to time (Uçar and Gölbaşı, 2015). In addition, pregnancy is a period in which biological, physiological and psychological changes occur in women. In pregnancy, which is a biologically normal process, the woman and the fetus must adapt to this situation in order to protect their health. Although the person experiencing pregnancy is a woman from a physiological point of view, close individuals around the pregnant woman are also involved in the process. In addition to the physiological and psychological changes that occur in the pregnant woman during pregnancy, the pregnant woman's spouse and other family members also experience some psychological and social changes and they need to adapt to these changes (Polat Başpınar, 2021).

The emotional state caused by these changes and the methods of coping with them vary from pregnant to pregnant. While most pregnant women can adapt to these situations brought about by pregnancy, many of them may experience serious problems during this period (Fırat, 2024). Various factors affect women's ability and ability to adapt to changes and challenges in pregnancy. These factors can be classified as personal, social, and pregnancy-related factors (Rockliffe et al., 2021).

Traditional and complementary medicine practices are used to reduce stress during pregnancy, to manage the discomfort experienced during pregnancy and to facilitate the adaptation process. It is increasing in popularity due to the fact that the vast majority of these methods are non-invasive and the awareness of the body-mind-spirit connection in health (Ağapınar Şahin and Bekar, 2023). Massage therapy, acupuncture, relaxation, yoga, homeopathy and aromatherapy are frequently used TTU methods to reduce stress and anxiety during pregnancy. Yoga is a nonpharmacological method that has become very popular recently, which is defined as a mental journey of the individual to his inner world. It reduces the stress caused by pregnancy and helps to reach a more peaceful and fulfilling life. It enables the mother to accept and connect to her body and baby (Şen et al. 2020).

Laughter yoga is an exercise that combines laughter and yoga breathing techniques. In addition, laughter yoga; It is a combination of relaxation technique, flexibility, aerobic exercise, and social interaction (Ağapınar Şahin and Bekar, 2022). Anyone can laugh without humor, jokes, comedy. Laughter sessions are done in a group, in the form of body exercises (Kataria, 2011). Those in the laughter group; As you maintain eye contact and childlike play, the laughter soon becomes real and contagious. In laughter yoga, the prevailing view is that the brain cannot distinguish between real and fake laughter. There is an argument that similar effects will be obtained because the brain cannot make this distinction (Kataria, 2011). Laughter yoga, which is used as a complementary and preventive treatment; Similar to traditional yoga, it is an exercise in which laughter is added to breathing, yoga and stress relief techniques. Laughter has physiological effects such as relaxing muscles, regulating breathing, stimulating circulation, increasing pain threshold and tolerance, reducing stress hormones such as cortisol and epinephrine, increasing the number of antibody-producing cells, and increasing the effectiveness of T cells (Tremayne and Sharma, 2019).

Pilates activates all muscle functions of the body and increases the endurance, flexibility and strength of all body muscles, especially the core area. Pilates is an exercise system that aims to improve dynamic postural control while improving the body's balance system (Srivastava, 2016). Pilates during pregnancy is one of the safe exercise methods that prepares and strengthens expectant mothers for childbirth from the first to the last month of pregnancy. Pilates can be done at least two or three times a week from the onset of pregnancy (Dillard, 2013). Regular exercises performed by the expectant mother play an important role in maintaining the psychological well-being of the mother during pregnancy. Internationally, Pilates is considered an important exercise to improve physical, psychological and motor functions. It supports the protection of self-esteem, self-efficacy and autonomy, a positive pregnancy and easy adaptation to motherhood (WHO, 2016). When examined in the literature, it has been reported that Pilates exercises performed regularly during pregnancy not only have a positive effect on pregnancy complaints and quality of life during pregnancy, but also increase stress management, decrease depression rates, low anxiety levels, and increase self-esteem and body image of pregnant women who exercise regularly (Aktan et al., 2021; Ghandali et al., 2021; Mazzarino et al., 2018). As a result, the aim of the study was to determine the effects of laughter yoga and pilates on pregnancy adjustment, anxiety and prenatal attachment in pregnant women who received childbirth preparation training.

ELIGIBILITY:
Inclusion Criteria:

Week of pregnancy over 20 weeks Without multiple and risky pregnancies, Those who have not undergone intra-abdominal surgery, Not having a mental illness, No physical disability, Without any fetal anomalies and intrauterine growth retardation, Pregnant women who agreed to participate in the study were included in the study.

Exclusion Criteria:

Incomplete filling of data forms, Not volunteering to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Pregnancy-Related Anxiety Scale | four week
  It is a 4-point Likert type scale consisting of a total of 33 questions. The scale consists of 9 sub-dimensions. In the scale, 11 items are reverse-coded, and the lowest score is 33 and the highest is 132 points.
Prenatal Self-Assessment Scale | four week
  It is a 4-point Likert-type scale consisting of 79 items. A minimum of 79 and a maximum of 316 points can be obtained on the scale
Prenatal Attachment Inventory | four week
  It consists of 21 items. Each item is of the quadruple Likert type, which can score between 1 and 4. A minimum of 21 and a maximum of 84 points can be obtained from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Demet Güney, MSc., Study Director — https://kastamonueah.saglik.gov.tr/
Locations (1):
- Demet Güney, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aktan B, Kayikcioglu F, Akbayrak T. The comparison of the effects of clinical Pilates exercises with and without childbirth training on pregnancy and birth results. Int J Clin Pract. 2021 Oct;75(10):e14516. doi: 10.1111/ijcp.14516. Epub 2021 Jul 5. PMID 34117824
- [Background] Baghdari N, Sadeghi Sahebzad E, Kheirkhah M, Azmoude E. The Effects of Pregnancy-Adaptation Training on Maternal-Fetal Attachment and Adaptation in Pregnant Women With a History of Baby Loss. Nurs Midwifery Stud. 2016 May 21;5(2):e28949. doi: 10.17795/nmsjournal28949. eCollection 2016 Jun. PMID 27556052
- [Background] Ghandali NY, Iravani M, Habibi A, Cheraghian B. The effectiveness of a Pilates exercise program during pregnancy on childbirth outcomes: a randomised controlled clinical trial. BMC Pregnancy Childbirth. 2021 Jul 2;21(1):480. doi: 10.1186/s12884-021-03922-2. PMID 34215198
- [Background] Mazzarino M, Kerr D, Morris ME. Pilates program design and health benefits for pregnant women: A practitioners' survey. J Bodyw Mov Ther. 2018 Apr;22(2):411-417. doi: 10.1016/j.jbmt.2017.05.015. Epub 2017 May 31. PMID 29861243
- [Background] Rockliffe L, Peters S, Heazell AEP, Smith DM. Factors influencing health behaviour change during pregnancy: a systematic review and meta-synthesis. Health Psychol Rev. 2021 Dec;15(4):613-632. doi: 10.1080/17437199.2021.1938632. Epub 2021 Jun 29. PMID 34092185
- [Result] Agapinar Sahin S, Bekar M. The influence of laughter yoga on pregnancy symptoms, mental well-being, and prenatal attachment: A randomized controlled study. Health Care Women Int. 2023 Jun;44(6):782-801. doi: 10.1080/07399332.2022.2164284. Epub 2023 Jan 10. PMID 36625775